CLINICAL TRIAL: NCT06399432
Title: Mediterranean Diet vs no Dietary Intervention for Improving Signs and Symptoms of Psoriasis in Patients Treated With Anti-IL-17 or Anti-IL-23 Inhibitors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Neil Korman, Principle Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20220312
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
Keywords: risankizumab; tildrakizumab; brodalumab; izekizumab; secukinumab; guselkumab
MeSH Terms: conditions — Psoriasis | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Active Comparator): Participants in this arm will follow the Mediterranean Diet.
  Interventions: Behavioral: Mediterranean Diet
- No Dietary Intervention (No Intervention): Participants in this arm will have no dietary intervention.

INTERVENTIONS:
Behavioral: Mediterranean Diet — In the Mediterranean Diet, all foods are included. Red meat will be limited to 1/week, poultry to ≤3 times/week and fish to 2-3 times/week. Supplementation with extra-virgin olive oil and nuts, providing 1 liter of olive oil per week and 30 gr a day of nuts.
  The dietician will personalize the dietary advice by adapting it to the patient's condition, preferences and beliefs, will encourage adherence, and transmit a sense of empowerment. A change in diet with specific, attainable goals will be negotiated between the dietician and the participant.
  Dieticians will conduct a phone call once in every 2-week period to assess dietary compliance using a 24-hour food recall, the Mediterranean Diet Adherence Form. MD patients will keep a diet diary for 3 days every two weeks, which they will discuss with the dietician during their scheduled dietician assessment. The Baseline Visit with the dietician can occur either in-person or via video communication software.
  Arms: Mediterranean Diet

SUMMARY:
In this study, participants will have 3 or 4 total study visits over approximately 10 total weeks. There is a two week medication washout period in between the 1st and 2nd visits. This washout only applies if participants are using a prohibited psoriasis medication (such as topical steroids or oral psoriasis medications, like methotrexate). During the washout period, participants will have to stop the prohibited medication(s). If participants are not using any prohibited medications, then the 1st and 2nd visits can be combined and participants will only have 3 total in-person visits. Participants will be randomly assigned (by chance; like flipping a coin) to either the Mediterranean Diet or no dietary intervention. After 4 weeks on the diet, participants will start treatment with either Anti-IL-17 or Anti-IL-23 therapy. The biologic treatments will prescribed by the participants regular dermatologist and not as a part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic plaque psoriasis for at least 12 months prior to Screening.
* Have moderate to severe plaque psoriasis at Baseline as defined by

  1. BSA ≥5% OR
  2. sPGA ≥3 (moderate to severe) OR
  3. PASI ≥5
* Must have been prescribed, per standard-of-care, an Anti-IL-17 or Anti-IL-23 therapy for psoriasis, which the patient has not yet started, but is willing to start during the study.

Eligible therapies are Secukinumab, Ixekizumab, Brodalumab, Guselkumab, Risankizumab, and Tildrakizumab.

* Must be in good health (except for psoriasis) as judged by the Investigator, based on medical history and physical examination.
* Must be eligible for a weight loss program, defined as being in good general health and having a BMI between 25 to 40.

Exclusion Criteria:

* Other than psoriasis, history of any clinically significant (as determined by the Investigator) cardiac (clinically advanced cardiovascular disease including stent, past history of MI, thrombotic event or arterial calcification), active or history of inflammatory bowel disease, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major uncontrolled disease.
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
* Any condition, including other inflammatory diseases or dermatologic conditions that confound the ability to interpret data from the study.
* Prior history of suicide attempt at any time in the subject's lifetime prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Pregnant or breast-feeding.
* Have failed more than 3 systemic agents for treatment of psoriasis.
* History of allergy to any component of Anti-IL-17 or Anti-IL-23 therapies.
* Had a serious infection (including, but not limited to, hepatitis, pneumonia, sepsis, cellulitis, meningitis or pyelonephritis) or have been hospitalized for an infection. Subject must be cured of infection > 4 weeks before Screening.
* Have a history of, or ongoing, chronic or recurrent infectious disease, including, but not limited to, chronic renal infection, chronic chest infection (e.g., bronchiectasis), sinusitis, recurrent urinary tract infection (e.g., recurrent pyelonephritis, chronic non-remitting cystitis), an open, draining, or infected skin wound or ulcer.
* Had a Bacillus Calmette-Guérin (BCG) vaccination within 1 year prior to screening.
* History of positive human immunodeficiency virus (HIV), or have congenital or acquired immunodeficiency (e.g., common variable immunodeficiency disease).
* Active substance abuse or a history of substance abuse within 6 months prior to Screening.
* Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment and cure for such infections must have been completed at least 4 weeks prior to Screening.
* Malignancy or history of malignancy, except for:

  1. treated [i.e., cured] basal cell or squamous cell in situ skin carcinomas;
  2. treated [i.e., cured] cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years.
* Have a known nut allergy.
* Currently participating in a supervised dietary program.
* Use of psoriasis therapy 2 weeks prior to Baseline (including, but not limited to, topical corticosteroids, retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, anthralin/dithranol, cyclosporine, corticosteroids, methotrexate, retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, sulfasalazine, azathioprine, fumaric acid esters, TNF inhibitors IL-17 inhibitors, IL-12/23 inhibitors, or phototherapy).

Exceptions: Low-potency corticosteroids will be allowed as background therapy and restricted to treatment of the face, axillae, and groin in accordance with the manufacturers' suggested usage during the course of the study (this restricted usage should be documented). Subjects with scalp psoriasis will be permitted to use coal tar shampoo and/or salicylic acid scalp preparations on scalp lesions. An unmedicated skin moisturizer (e.g. Eucerin®) will be also permitted for body lesions only. Subjects should not use these topical treatments within 24 hours prior to the clinic visit.

* Use of any investigational drug within 2 weeks prior to Baseline.
* Prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources.
* Currently flaring or unstable psoriasis.

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who had a change in blood monocytes profiles. | Baseline, 10 weeks
Percentage of participants who had a change in T-cell profiles. | Baseline, 10 weeks
Change in blood monocyte profile. | Baseline, 10 weeks
Change in T-cell profiles. | Baseline, 10 weeks

SECONDARY OUTCOMES:
Change in serum biomarkers. | Baseline, 10 weeks
Change in gut microbiome. | Baseline, 10 weeks
Change in single cell gene expression. | Baseline, 10 weeks
Change in metabolomics profile. | Baseline, 10 weeks
Change in serum chemistries. | Baseline, 10 weeks
Change in complete blood cell count. | Baseline, 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil Korman, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Jordan K Kahle, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No